CLINICAL TRIAL: NCT06635915
Title: Ultrasound to Check the Adequate Position of the Nasogastric Tube to Improve Patient Management and Safety
Brief Title: Ultrasound to Check the Position of the Nasogastric Tube
Acronym: SONUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Negrin University Hospital (Other)
Responsible Party: Principal Investigator, Ángel Becerra, Principal Investigator, Dr. Negrin University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2022-300-1
Record Dates: First submitted 2024-10-07; First posted 2024-10-10 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Nasogastric Tube Placement
Keywords: nasogastric tube placement; ultrasound; postoperative diagnosis; monitoring

STUDY DESIGN:
Intervention Model Description: Clinical trial that will include patients who have had NGT placed intraoperatively. 114 patients (57 with NGT and 57 without NGT) will be examined by ultrasound in the immediate postoperative period to diagnose the normal positioning of the NGT or its absence. In patients who have had NGT placed, the normal positioning of the NGT will be verified by chest X-ray.
Who Masked: Care Provider, Investigator
Masking Description: The upper part of the patients will be covered for the investigator, who will only have access to the patient's abdomen and will not know which patients have NGT or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with nasogastric tube placed during the intraoperative period. (Experimental): Ultrasound will be performed during the postoperative period to assess the normoposition of nasogastric tube.
  Interventions: Diagnostic Test: Postoperative ultrasound
- Patients without nasogastric tube placed during the intraoperative period. (Active Comparator): Ultrasound will be performed during the postoperative period to assess the absence of nasogastric tube.
  Interventions: Diagnostic Test: Postoperative ultrasound

INTERVENTIONS:
Diagnostic Test: Postoperative ultrasound — Ultrasound will be performed to both groups in the postoperative period to assess the normoposition or the absence of nasogastric tube.

SUMMARY:
The main objective of this study is to evaluate whether the use of ultrasound as a method of checking the normal positioning of the NGT is reliable, without requiring other diagnostic tests. Clinical trial that will include patients who had the NGT placed intraoperatively. 114 patients (57 with NGT and 57 without NGT) will be examined by ultrasound in the immediate postoperative period to diagnose the normal positioning of the NGT or its absence.

Can ultrasound quickly and effectively diagnose the normal positioning of the NGT? Can chest X-ray be avoided by introducing ultrasound in the verification of the normal positioning of the NGT in the immediate postoperative period?

DETAILED DESCRIPTION:
The nasogastric tube (NGT) is an essential element of our daily clinical practice, commonly used for the administration of enteral nutrition and medication or for gastric decompression and diagnostic procedures. Despite its common use, it is still an invasive procedure with potential complications. Ultrasound is a noninvasive, inexpensive, widely available and rapid method that can speed up the proper verification of these devices. The main objective of this study is to evaluate whether the use of ultrasound as a method of checking the normal positioning of the NGT is reliable, without requiring other diagnostic tests. Clinical trial that will include patients who had the NGT placed intraoperatively. 114 patients (57 with NGT and 57 without NGT) will be examined by ultrasound in the immediate postoperative period to diagnose the normal positioning of the NGT or its absence. Patients who have had the NGT placed will have had their NGT placed correctly by chest X-ray. The upper part of the patient will be covered for the examiner, who will only have access to the patient's abdomen and will not know which patients have NGT or not.

ELIGIBILITY:
Inclusion Criteria:

* Patients classified as ASA I-IV according to the American Society of Anesthesiologists
* Patients over 18 years old.
* Informed consent signed by the patient or their family representatives

Exclusion Criteria:

* Patients classified as ASA V.
* Patients under 18 years old.
* Refusal to participate in the study.
* Contraindication for nasogastric tube placement: ingestion of caustics, nasal or skull fractures, and cervical surgery.
* Patients with anatomical abnormalities at the cervical or pharyngoesophageal level.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Rate of confirmation of normoposition of the nasogastric tube | First postoperative hour.
  Researchers will perform postoperative abdominal ultrasound to verify proper placement of the nasogastric tube in patients who have one or its absence in those who have not had one.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario de Gran Canaria Doctor Negrín, Palmas de GRAN Canaria, LAS, Las Palmas
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria

IPD SHARING:
Plan to Share IPD: Undecided